CLINICAL TRIAL: NCT04958616
Title: Association Between House Dust Mites Sensitization and Level of Asthma Control and Severity in Children Attending Mansoura University Children's Hospital.
Brief Title: House Dust Mites Sensitization and Level of Asthma Control and Severity in Children
Status: Completed | Type: Observational
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Engy Osman Ahmed, Assistant professor of pediatrics, allergy and clinical immunology unit., Mansoura University Children Hospital
Other Study IDs: Ms.18.07.201
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Bronchial Asthma
Keywords: Asthma severity; House dust mites.
MeSH Terms: conditions — Asthma | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample was collected in EDTA tube for assessment of Eosinophil count and Serum IgE.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients sensitive to HDM: Classification of asthma according to disease severity. Patient maintained on step 2 treatments are often classified as having mild asthma. Those receive step 3-4 as moderate asthma and those prescribed step 4-5 as having moderate to severe asthma. Assessment level of asthma control Based on asthma control score according to GINA guideline defined as controlled, partially controlled and well controlled.Skin prick test: for (Dermatophagoides pteronyssinus and Dermatophagoides Farina). Through the use of specific allergen extracts, positive and negative controls, then interpretation after 15-20 minutes of maneuver, a wheal ≥3 mm diameter is considered positive [9]. Before the test, we checked that the patient has not taken medications that might interfere with the test and antihistamines had stopped using before the skin prick test (2 days for the first generation and 7 days for the second generation)
  Interventions: Diagnostic Test: Skin prick test.
- Patients not sensitive to HDM allergy.: Classification of asthma according to disease severity. Patient maintained on step 2 treatments are often classified as having mild asthma. Those receive step 3-4 as moderate asthma and those prescribed step 4-5 as having moderate to severe asthma. Assessment level of asthma control Based on asthma control score according to GINA guideline defined as controlled, partially controlled and well controlled .Skin prick test: for (Dermatophagoides pteronyssinus and Dermatophagoides Farina). Through the use of specific allergen extracts, positive and negative controls, then interpretation after 15-20 minutes of maneuver, a wheal ≥3 mm diameter is considered positive [9]. Before the test, we checked that the patient has not taken medications that might interfere with the test and antihistamines had stopped using before the skin prick test (2 days for the first generation and 7 days for the second generation).
  Interventions: Diagnostic Test: Skin prick test.

INTERVENTIONS:
Diagnostic Test: Skin prick test. — Skin prick test: for (Dermatophagoides pteronyssinus and Dermatophagoides Farina). Through the use of specific allergen extracts, positive and negative controls, then interpretation after 15-20 minutes of maneuver, a wheal ≥3 mm diameter is considered positive [9]. Before the test, we checked that the patient has not taken medications that might interfere with the test and antihistamines had stopped using before the skin prick test (2 days for the first generation and 7 days for the second generation)
  Other Names: pulmonary function tests ,spirometry.

SUMMARY:
In this study we aimed to assess the clinical and laboratory profile of some Egyptian asthmatic children who are sensitized to house dust mites and determine the association of HDM sensitization and severity of asthma according to recent GINA guidelines.

DETAILED DESCRIPTION:
This is an observational, case control study. The study was carried out in Allergy, Clinical Immunology and pediatric pulmonology Unit; at Mansoura University Children Unit during the years 2018-2019. The study included 60 children above 6 years with atopic asthma. They were 42 males and 18 females, their age ranged from 8-17 years. Bronchial asthma diagnosis was based on clinical manifestations and spirometry results. Atopy was defined as presence of symptoms of atopic dermatitis, allergic rhino conjunctivitis, or food allergy, it was confirmed when asthmatic children fulfilled one of the following criteria: higher serum level of total IgE (more than 32IU/ml), eosinophilia (differential count more than 5% or absolute count more than 450/µl) or positive skin prick test (3 mm greater than control).

Asthmatic children were maintained on controller therapy for at least 6 months. They were classified according to skin prick test results into two groups:

* Group1: It included 30 atopic asthmatic children, who were sensitive to one of the two HDM (D pteronyssinus or D farina).
* Group2: It included 30 atopic asthmatic children who were not sensitive to HDM allergy.
* Sampling Samples were convenient and patients were enrolled in the study by consecutive manner.

history taking

* Personal and demographic data e.g. age, sex and residence.
* Asthma symptoms; cough, wheeze, as well as exercise-induced asthma.
* Symptoms of other atopic diseases in the child including allergic march.
* Based on frequency of each symptom, assessment of asthma control was done according to GINA 2017.

Pulmonary Function Test (Spirometry) Forced expiratory volume in 1 second FEV1%; forced vital capacity (FVC %); FEV1/FVC ratio and forced expiratory flow rate from 25% to 75% of vital capacity (FEF25-75%) were measured by spirometry (Master Screen pediatrics). The highest reading of three successive measurements was taken. Reference values were computed according to the recommendations of the American Thoracic Society standards of acceptability and reproducibility in subjects above the age of 6 years who need cooperation for forced respiratory maneuver.

Skin prick test: for (Dermatophagoides pteronyssinus and Dermatophagoides Farina). Through the use of specific allergen extracts, positive and negative controls, then interpretation after 15-20 minutes of maneuver, a wheal ≥3 mm diameter is considered positive. Before the test, we checked that the patient has not taken medications that might interfere with the test and antihistamines had stopped using before the skin prick test (2 days for the first generation and 7 days for the second generation).

3- Eosinophil count Blood sample was collected in EDTA tube. Total leucocytic count and eosinophilia % were determined by automated cell counter [11].

4- Serum IgE Blood samples were collected into tubes with ethylene tetr-acetic acid (EDTA). After incubation at room temperature for 20 minutes, tubes were centrifuged for 15 minute at 2500 revolutions per minute (rpm). Supernatant levels of IgE were determined by the ELISA technique [12].

Assessment level of asthma severity Classification of asthma according to disease severity is defined level (mild, moderate, severe) according to treatment steps when the patient has been maintained on regular controller therapy for several months. Patient maintained on step 2 treatments are often classified as having mild asthma. Those receive step 3-4 as moderate asthma and those prescribed step 4-5 as having moderate to severe asthma [2].

I) Assessment level of asthma control based on asthma control score according to GINA guideline defined as controlled, partially controlled and well controlled .

Statistical analysis

Data were fed to the computer and analyzed using IBM SPSS Corp. Released 2013. IBM SPSS Statistics for Windows, Version 22.0. Armonk, NY: IBM Corp. The following tests were used:

Qualitative data: Chi-Square test for comparison of 2 or more groups. Monte Carlo test as correction for Chi-Square test when more than 25% of cells have count less than 5 in tables (>2*2).

ELIGIBILITY:
Inclusion Criteria:

* Age more than 6 years.
* Asthmatic children with history of atopy (atopic dermatitis, allergic rhinitis or food allergy).

Exclusion Criteria:

* Other diseases which influence bronchial symptoms and/or lung function.
* Patients weren't compliant with asthma therapy.
* Refused the informed consent.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study was carried out in Allergy, Clinical Immunology and pediatric pulmonology Unit; at Mansoura University Children hospital.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Assessment of asthma severity and level of control. | 1 year
  . Patient maintained on step 2 treatments are often classified as having mild asthma. Those receive step 3-4 as moderate asthma and those prescribed step 4-5 as having moderate to severe asthma. Based on asthma control score according to GINA guideline defined as controlled, partially controlled and well controlled

CONTACTS AND LOCATIONS:
Locations (1):
- Amr Sarhan, Al Mansurah, None Selected, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Global Initiative for Asthma. Global Strategy for Asthma Management and Prevention, 2020 — https://ginasthma.org/?fbclid=IwAR1EKFqnZgdkBtjoLP2J1O_Uyk6GhfzdWEbNSbWJHTPrNKIZ-vBXan2AJD4